CLINICAL TRIAL: NCT02278926
Title: Ultrasound Characterization of Lipo-hypertrophy in Type 1 Diabetes Mellitus
Brief Title: Lypo-hypertrofia Characterization in Diabetes
Status: Completed | Type: Observational
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 442-092014
Record Dates: First submitted 2014-10-27; First posted 2014-10-30 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Ultrasound; Lypo-hypertrophy
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients ultrasound lypo-hypertrophy identification: Type 1 diabetes patients with visible lypo-hypertrphy attended in outpatient clinic
  Interventions: Other: Ultrasound
- Control group: Type 1 diabetes patients with visible lypo-hypertrphy attended in outpatient clinic
  Interventions: Other: Tapping and body inspection to define the area of insulin injection

INTERVENTIONS:
Other: Ultrasound — Ultrasound measurements
  Groups: Patients ultrasound lypo-hypertrophy identification
Other: Tapping and body inspection to define the area of insulin injection — Obese patients with a thickening fat subcutaneous tissue that could have interfered with the interpreting and analyzing of the data are left out of this first study. In the control group we manage to define the lypo-hypertrophic area by tapping and body inspection
  Groups: Control group

SUMMARY:
Aim/hypothesis: Subcutaneous insulin absorption is one of the factors which strongly influence blood sugar control in patients with diabetes mellitus on insulin therapy. In response, a regular absorption is influenced by lipo-hypertrophy in subcutaneous tissue on injection sites. So far lipo-hypertrophy diagnosis has only been clinical since there are no imaging studies that have characterized precisely morphometry of lipo-hypertrophic tissue. Methods: In two groups of 20 type 1 diabetes patients on insulin therapy, lipo-hypertrophy is characterized and defined by clinical tapping or by ultrasound with multi frequency linear probe (6-18 Mhz). Patients are therefore advised to avoid insulin injections on those areas so defined. Patients are reevaluated 3 and 12 months later

DETAILED DESCRIPTION:
An observational study has been carried out, checked with parallel arms in which type 1 diabetes patients are recruited with clinical evidence of lypo-hypertrophy in insulin injected areas. Patients attend to the Diabetes Unit of Niguarda Ca' Granda Hospital. Obese patients with a thickening fat subcutaneous tissue that could have interfered with the interpreting and analyzing of the data are left out of this first study. In the control group the investigators manage to define the lypo-hypertrophic area by tapping and body inspection. In the study group the investigators can define and mark out the area/areas with lipo-hypertrophy by ultrasound scan test. All the tested patients both the control group and the study group, are discouraged from use insulin in areas where lypo-hypertrophy is present. Patients are reassessed after 3 months with a clinical assessment of glucose control by HbA1c. After 12 months subcutaneous tissue scan is repeated in 10 patients within the experimental group and a new assessment of HbA1c is performed. Ultrasound assessment. The scan used is Esaote My Lab70 linear probe multi-frequency [6-18 Mhz)

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes
* age between 18 and 75 years old
* lack of extended cutaneous diseases
* BMI <30

Exclusion Criteria:

* BMI> 30
* active allergies
* cancer
* liver failure
* kidney failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type 1 diabetes patients with visible lypo-hypertrphy that attend consecutively in our outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Glucose control | month 3
  Glucose control by insulin therapy, measured by HbA1c values

SECONDARY OUTCOMES:
Glucose control | month 12
  Glucose control by insulin therapy, measured by HbA1c values

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Bruschi, MD, Study Chair — Niguarda Hospital; Oscar Epis, MD, Study Chair — Niguarda Hospital; Federico Bertuzzi, MD, Principal Investigator — Niguarda Hospital
Locations (1):
- Nigurada Hospital, Milan, Italy